CLINICAL TRIAL: NCT05901077
Title: European Cystinosis Cohort
Acronym: RaDiCo-ECYSCO
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-49
Record Dates: First submitted 2022-03-11; First posted 2023-06-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cystinosis
Keywords: Quality of life; Effects of treatments; European Study
MeSH Terms: conditions — Cystinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystinosis is a generalized lysosomal storage disease with a reported incidence of about 1:180,000 live births. There are estimated 110-140 cases in France (approximately 500 in Western Europe). The disease is caused by mutations in the CTNS gene coding for cystinosin, a lysosomal carrier protein. The lysosomal cystine accumulation leads to cellular dysfunction in many organs. The first symptoms start at about 6 months of age. In the absence of specific therapy, end stage renal disease occurs between 6 and 12 years of age. Survival beyond this age is associated with the development of extra-renal complications.

Renal transplantation and the availability of cystine-depleting medical therapy, cysteamine (EU/1/97/039/001, EU/1/97/039/003), have radically altered the natural history of cystinosis. Cystinosis is a good example of a "paediatric" disease where patients now survive into adolescence and adulthood. These individuals have complex, multisystem problems that require on-going care.

Despite some progress in recent years there are still significant limitations in the knowledge of diagnostic and therapeutic procedures. A first European registry was launched in 2011, using the CEMARA application developed by the Banque Nationale de Données Maladies Rares (BNDMR, CNIL authorisation number: 1187326), allowing the collection of data from France, Belgium and Italy. The objective of the current study is to translate this database into a cohort study that will allow and facilitate the collection of a wider range of data including clinical, and personal data such as quality of life data, from an increased number of European countries, improve the monitoring, data-management and analysis of the data, offer the possibility for patients to actively participate to and benefit from the study by developing a module in which patients will enter their own data on quality of life with a direct feed-back on the general results.

This project is a unique opportunity for building a consensual European academic cohort not based on company driven, "drug-oriented" objectives.

The cohort will collect clinical details to analyse patient outcomes thus providing audit of patient care & clinical effectiveness. It will be possible, through the cohort, to indicate where improvements need to be made and ultimately improve care to the highest standards.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystinosis (based on cystine dosage, presence of crystals at eye examination or molecular diagnosis)
* Signed informed consent

Exclusion Criteria:

* Patients not able to give their informed consent. No other criteria (patients with associated disease should be enrolled).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prevalent subjects will be selected in european country such as France, Belgium, Italy, Germany and Spain via the CEMARA registry.
  French paediatric patients suspected with cystinosis are first sent to a nephrologist who will redirect them to centres of reference/competence where the confirmation of the diagnosis will be performed either by cysteine dosage, presence of intra-ocular cysteine crystals detection and combined, when possible, by genetic analysis.
  For french patients who declared the disease once adult, the diagnosis is mainly made by ophthalmologist who identify the presence of ocular cysteine crystals.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in the number of renal replacement therapy (RRT) | Through study completion, at 1 year, 2 year, 3 year
Change in Estimated Glomerular Filtration Rate (eGRF) | Through study completion, at 1 year, 2 year, 3 year

SECONDARY OUTCOMES:
Endocrine manifestations | Through study completion, at 1 year, 2 year, 3 year
  * Tanner scale for pubertal and genital state,
  * Age of Menarche,
  * Presence of hypothyroidism,
  * Diabetes mellitus and impaired glucose tolerance
Memory loss, cognitive defect, speech disorder with a Questionnaires | Through study completion, at 1 year, 2 year, 3 year
Seizure, stroke, motor defect, extrapyramidal movement disorder reported from patients files | Through study completion, at 1 year, 2 year, 3 year
Sensory neuropathy, neuroradiological signs, somnolence, collected by the physicians during the visits | Through study completion, at 1 year, 2 year, 3 year
Treatment compliance | Through study completion, at 1 year, 2 year, 3 year
  Records of adverse events for the long-term safety of treatment (side effects of eye drops -presence of redness, blurring, irritation, itching, pain, or of skeletal, haematological, biochemical, etc. manifestations), treatment duration and interuption and treatment compliance records.
Genetics | At inclusion
  Description of mutations encountered within population in particular in CTNS gene (57Kb deletion and others mutations)

CONTACTS AND LOCATIONS:
Overall Officials: Aude Servais, PHD, Principal Investigator — INSERM U933
Locations (1):
- RaDiCo-ECYSCO, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided